CLINICAL TRIAL: NCT06265051
Title: Safety and Efficacy of Adjunct Tirofiban Treatment After Successful Mechanical Thrombectomy Recanalization in Acute Anterior Circulation Ischemic Stroke- A Multicenter, Prospective, Double-blind, Randomized Trial
Brief Title: Tirofiban After Successful MT Recanalization in AIS
Acronym: ATTRACTION
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiang Luo (Other)
Collaborators: Wuhan Central Hospital (Other); Zhongnan Hospital (Other); Renmin Hospital of Wuhan University (Other); Second Affiliated Hospital of Soochow University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Wuhan Hospital of Traditional Chinese Medicine (Other); The Central Hospital of Enshi Tujia And Miao Autonomous Prefecture (Other); Huangshi Central Hospital (Other); The First Affiliated Hospital of Yangtze University (Other); The Fifth Hospital of Wuhan (Other); Wuhan Puren Hospital (Other); Xiangyang No.1 People's Hospital (Other); Xianning Central Hospital (Other); Hanyang University (Other); Wuhan Third Hospital (Other); Yichang Central People's Hospital (Other); Affiliated Hospital of Chengde Medical University (Other); Beijing Tiantan Hospital (Other); Nanyang Central Hospital (Other); Jingzhou Central Hospital (Other); Taihe Hospital (Other); The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor-Investigator, Xiang Luo, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100939
Record Dates: First submitted 2024-02-09; First posted 2024-02-20 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke; Vessel Occlusion
Keywords: mechanical thrombectomy; acute ischemic stroke; successful recanalization; tirofiban
MeSH Terms: conditions — Ischemic Stroke | interventions — Tirofiban; Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tirofiban group (Experimental): After the completion of endovascular treatment and successful recanalization (mTICI 2b/3), the patients were randomly assigned to the experimental group. Tirofiban 5μg/kg was administered intravenously through the catheter artery at a rate of 1ml/min, followed by an intravenous infusion of 0.1μg/(kg·min) for 24 hours. Standard medical treatment was administered after the surgery.
  Interventions: Drug: Tirofiban
- placebo group (Placebo Comparator): After the completion of endovascular treatment and successful recanalization (mTICI 2b/3), the patients were randomly assigned to the control group. Saline placebo was administered in the same manner as tirofiban group. Standard medical treatment was administered after the surgery.
  Interventions: Drug: Saline placebo

INTERVENTIONS:
Drug: Tirofiban — After the completion of endovascular treatment and successful recanalization (mTICI 2b/3), the patients were randomly assigned to the experimental group. Tirofiban 5μg/kg was administered intravenously through the catheter artery at a rate of 1ml/min, followed by an intravenous infusion of 0.1μg/(kg·min) for 24 hours. Standard medical treatment was administered after the surgery.
  Other Names: trade name: Xinweining; Wuhan Grand Pharmaceutical Group Co., LTD. (China)
  Arms: Tirofiban group
Drug: Saline placebo — After the completion of endovascular treatment and successful recanalization (mTICI 2b/3), the patients were randomly assigned to the experimental group. Saline placebo was administered in the same manner as tirofiban group. Standard medical treatment was administered after the surgery.
  Arms: placebo group

SUMMARY:
Acute ischemic stroke with large vessel occlusion is a frequently occurring life-threatening condition. Although endovascular treatment can effectively open occluded vessels, the successful reperfusion rate exceeds 80%, but the rate of good prognosis is less than 50%. The current clinical focus is on how to improve futile recanalization. Tirofiban is widely used in the treatment of stroke, as it can effectively prevent vascular reocclusion and improve microcirculation perfusion. It has the potential to improve futile recanalization, but there is a lack of high-level evidence-based medical support. This multicenter, prospective, double-blind, randomized controlled trial was conducted to assess the effectiveness and safety of sequential tirofiban therapy following successful mechanical thrombectomy within 24 hours of onset.

DETAILED DESCRIPTION:
Endovascular treatment is the primary approach for significantly improving the clinical prognosis of patients with acute large vessel occlusion, and it has been consistently recommended by both domestic and foreign guidelines. Successful vascular recanalization and restoration of ischemic tissue reperfusion are crucial for the favorable prognosis of patients with large vessel occlusion. However, the rate of successful reperfusion after endovascular treatment exceeds 80%, but the rate of favorable outcomes at 90 days follow-up is less than 50%. The reasons for ineffective recanalization include reperfusion injury, arterial reocclusion, hemorrhagic transformation, and microvascular reperfusion insufficiency. Although vascular recanalization can be visualized using DSA, not all microvascular beds can be effectively perfused, and persistent microocclusion of the capillary bed in ischemic tissue will also result in a poor prognosis. Currently, drug intervention is not commonly utilized to achieve successful recanalization after mechanical thrombectomy in clinical practice. Additionally, there is a lack of effective methods to improve ineffective recanalization.

Tirofiban is widely used in the treatment of stroke, as it can effectively prevent vascular reocclusion and improve microcirculation perfusion. It has the potential to improve futile recanalization, but there is a lack of high-level evidence-based medical support.

This is a prospective, randomized, multicenter, double-blind clinical trial. In 52 centers in China, 1360 patients with the following situations will be enrolled: achieved successful recanalization after mechanical thrombectomy (mTICI 2b/3) within 24h of stroke onset.

Patients will be randomly assigned into 2 groups according to the ratio of 1:1:

1. experimental group received a bolus of tirofiban at a dosage of 5μg/kg (with a maximum dose not exceeding 0.5mg) through the catheter artery, followed by a continuous intravenous infusion at a rate of 0.1μg/(kg·min) for 24 hours.
2. The control group was given a placebo in the same manner. Face to face interviews will be made on baseline, 24 hours after randomization, 48 hours after randomization, day 7 after randomization or discharge day. Day 90 after randomization will be interviewed by phone or face to face.

The main measure of effectiveness was the rate of mRS 0-2 after 90 days, and the primary focus on safety was the rate of symptomatic intracranial hemorrhage within 48 hours. This study aims to clarify the role of tirofiban in enhancing unsuccessful recanalization after thrombectomy, which holds significant clinical value in improving the prognosis of patients following thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. NIHSS score: 6-30;
3. Symptom onset to random time of 24h, including wake-up stroke or unwitnessed stroke; The onset time of symptoms was defined as the last time of normal performance.
4. mRS 0-1 before the stroke;
5. Subject or legal representative can sign an informed consent form;
6. Clinical symptoms caused by acute occlusion of the following sites confirmed by CTA or MRA: intracranial segment of ICA, M1 segment of middle cerebral artery, M2 trunk of middle cerebral artery;
7. ASPECTS≥6 on NCCT or DWI;
8. After the end of mechanical thrombectomy, the mTICI was stable at 2b/3, and there was no secondary embolism in other non-offending vessels, or the diagnostic angiography before mechanical thrombectomy showed that the occluded vessels improved to mTICI 2b/3, and no mechanical thrombectomy was planned.

Exclusion Criteria:

1. Intra-arterial thrombolysis;
2. Tirofiban was used within 24 hours before endovascular treatment
3. Women who are known to be pregnant or lactating, or have a positive pregnancy test before randomization;
4. Allergy to tirofiban, radiocontrast agent or Nitinol materials;
5. Any active bleeding within 30 days before stroke or recent bleeding (gastrointestinal, urinary, etc.);
6. parenchymal organ surgery or biopsy within 14 days before stroke;
7. History of heparin-induced thrombocytopenia;
8. Platelet count < 100*10^9/L;
9. Being on hemodialysis or peritoneal dialysis; Known severe renal insufficiency (glomerular filtration rate < 30ml/min or serum creatinine > 220μmol/L).
10. Subjects requiring hemodialysis or peritoneal dialysis or who have contraindications to angiography for any reason;
11. The expected survival time is less than half a year (such as malignant tumors, serious heart and lung diseases, etc.);
12. Have participated in other interventional clinical studies that may have an impact on the outcome assessment;
13. Other circumstances that the investigator considers inappropriate for participation in the study or that may pose a significant risk to the patient (e.g., inability to understand and/or comply with study procedures and/or follow-up due to mental illness, cognitive or emotional disorder).
14. The midline shift of the brain or cerebral hernia, ventricular mass effect;
15. Acute intracranial hemorrhage on CT or MRI;
16. New bilateral acute stroke or intracranial multi-drainage large vessel occlusion;
17. Simple extracranial occlusion of the internal carotid artery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1380 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2025-12-29 (Actual); Study Completion 2025-12-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients functionally independent (mRS score 0 to 2) at 90 days | 90 days after randomization
  independent outcome at 90 days
Number of participants with symptomatic intracranial hemorrhage | within 48 hours of randomization
  According to Heidelberg Bleeding Classification

SECONDARY OUTCOMES:
Modified ranking scale (mRS) | 90 days after randomization
  A 0-6 scale running from perfect health without symptoms to death
Proportion of patients non-disabled (mRS score 0 to 1) or return to pre-morbid mRS score at 90 days (for patients with mRS > 1) | 90 days after randomization
  Excellent functional outcome
Proportion of patients ambulatory or bodily needs-capable or better (mRS score 0 to 3) | 90 days after randomization
  Ambulatory or bodily needs-capable or better
Number of participants with improvement of neurological function | 36 hours (24-48 hours) after randomization
  Proportion of patients with an NIHSS score of 0-1 or a reduction of ≥4 points from baseline at 36 hours (24-48 hours) of randomization
Health-related quality of life, assessed with the European Quality Five Dimensions Five Level scale (EQ-5D-5L) | 90 days after randomization
  Health-related quality of life
All-cause mortality | 90 days after randomization
  The ratio of total deaths from all causes to the research subjects at 90 days of randomization
Proportion of intracranial hemorrhage of any type | within 48 hours of randomization
  Proportion of intracranial hemorrhage of any type within 48 hours of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Luo, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renu A, Millan M, San Roman L, Blasco J, Marti-Fabregas J, Terceno M, Amaro S, Serena J, Urra X, Laredo C, Barranco R, Camps-Renom P, Zarco F, Oleaga L, Cardona P, Castano C, Macho J, Cuadrado-Godia E, Vivas E, Lopez-Rueda A, Guimaraens L, Ramos-Pachon A, Roquer J, Muchada M, Tomasello A, Davalos A, Torres F, Chamorro A; CHOICE Investigators. Effect of Intra-arterial Alteplase vs Placebo Following Successful Thrombectomy on Functional Outcomes in Patients With Large Vessel Occlusion Acute Ischemic Stroke: The CHOICE Randomized Clinical Trial. JAMA. 2022 Mar 1;327(9):826-835. doi: 10.1001/jama.2022.1645. PMID 35143603
- [Background] Dornbos D 3rd, Katz JS, Youssef P, Powers CJ, Nimjee SM. Glycoprotein IIb/IIIa Inhibitors in Prevention and Rescue Treatment of Thromboembolic Complications During Endovascular Embolization of Intracranial Aneurysms. Neurosurgery. 2018 Mar 1;82(3):268-277. doi: 10.1093/neuros/nyx170. PMID 28472526
- [Background] Guan Q, Yun W, Li X, Ni H, Lv W, Xie Z, Zhang L, Zhou J, Xu Y, Li J, Zhang Q. Association of tirofiban with improvement of functional outcomes of direct thrombectomy for acute anterior circulation occlusion: a retrospective, nonrandomized, multicenter, real-world study. Neurosurg Focus. 2023 Oct;55(4):E21. doi: 10.3171/2023.7.FOCUS23150. PMID 37778035
- [Background] RESCUE BT Trial Investigators; Qiu Z, Li F, Sang H, Luo W, Liu S, Liu W, Guo Z, Li H, Sun D, Huang W, Zhang M, Zhang M, Dai W, Zhou P, Deng W, Zhou Z, Huang X, Lei B, Li J, Yuan Z, Song B, Miao J, Liu S, Jin Z, Zeng G, Zeng H, Yuan J, Wen C, Yu Y, Yuan G, Wu J, Long C, Luo J, Tian Z, Zheng C, Hu Z, Wang S, Wang T, Qi L, Li R, Wan Y, Ke Y, Wu Y, Zhu X, Kong W, Huang J, Peng D, Chang M, Ge H, Shi Z, Yan Z, Du J, Jin Y, Ju D, Huang C, Hong Y, Liu T, Zhao W, Wang J, Zheng B, Wang L, Liu S, Luo X, Luo S, Xu X, Hu J, Pu J, Chen S, Sun Y, Jiang S, Wei L, Fu X, Bai Y, Yang S, Hu W, Zhang G, Pan C, Zhang S, Wang Y, Cao W, Yang S, Zhang J, Guo F, Wen H, Zhang J, Song J, Yue C, Li L, Wu D, Tian Y, Yang J, Lu M, Saver JL, Nogueira RG, Zi W, Yang Q. Effect of Intravenous Tirofiban vs Placebo Before Endovascular Thrombectomy on Functional Outcomes in Large Vessel Occlusion Stroke: The RESCUE BT Randomized Clinical Trial. JAMA. 2022 Aug 9;328(6):543-553. doi: 10.1001/jama.2022.12584. PMID 35943471
- [Background] Zhong HL, Zhou TF, He YK, Li TX, Li ZS. Safety and efficacy of adjunct tirofiban treatment following mechanical thrombectomy for acute ischemic stroke patients with large vessel occlusion (LVO) resulting in successful reperfusion. Interv Neuroradiol. 2024 Oct;30(5):657-662. doi: 10.1177/15910199221138883. Epub 2022 Nov 10. PMID 36358016